CLINICAL TRIAL: NCT04314843
Title: A Phase 1/2 Open-label, Multicenter Study of Lenzilumab and Axicabtagene Ciloleucel in Subjects With Relapsed or Refractory Large B-cell Lymphoma (ZUMA-19)
Brief Title: Study of Lenzilumab and Axicabtagene Ciloleucel in Participants With Relapsed or Refractory Large B-Cell Lymphoma
Acronym: ZUMA-19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Development program terminated and the decision was not due to any safety concerns.
Sponsor: Kite, A Gilead Company (Industry)
Collaborators: Humanigen, Inc. (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KT-US-471-0119; 2019-004568-23 (EudraCT Number)
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-07

CONDITIONS: Relapsed/Refractory Large B-cell Lymphoma
Keywords: Granulocyte Macrophage-Colony Stimulating Factor (GM-CSF); GM-CSF antibody; Chimeric Antigen Receptor (CAR); CD19
MeSH Terms: conditions — Recurrence | interventions — Cyclophosphamide; fludarabine; lenzilumab; axicabtagene ciloleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenzilumab and Axicabtagene Ciloleucel (Experimental): Phase 1: Participants will receive cyclophosphamide and fludarabine lymphodepleting chemotherapy followed by sequenced therapy of lenzilumab and axicabtagene ciloleucel on Day 0 to determine a recommended Phase 2 dose (RP2D) of lenzilumab. Phase 2: Participants will receive cyclophosphamide and fludarabine lymphodepleting chemotherapy followed by sequenced therapy of lenzilumab, at the RP2D, and axicabtagene ciloleucel on Day 0.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Lenzilumab; Biological: Axicabtagene Ciloleucel

INTERVENTIONS:
Drug: Cyclophosphamide — Administered according to package insert
Drug: Fludarabine — Administered according to package insert
Biological: Lenzilumab — Administered as an IV infusion
  Other Names: Humaneered® anti-human GM-CSF monoclonal antibody
Biological: Axicabtagene Ciloleucel — A single infusion of chimeric antigen receptor (CAR) transduced autologous T cells administered intravenously.
  Other Names: Yescarta®

SUMMARY:
The primary objectives of this study are:

Phase 1: To evaluate the safety of sequenced therapy with lenzilumab and axicabtagene ciloleucel in participants with relapsed or refractory large B-cell lymphoma and identify the most appropriate dose of lenzilumab for Phase 2.

Phase 2: To evaluate the incidence of neurologic events with sequenced therapy given at the recommended Phase 2 dose (RP2D) of lenzilumab in participants with relapsed or refractory large B-cell lymphoma.

DETAILED DESCRIPTION:
This study was intended to be a Phase 1/2, but the planned Phase 2 part has been canceled.

All participants who received an infusion of lenzilumab and axicabtagene ciloleucel will be provided the opportunity to transition to a separate long-term follow-up (LTFU) study, KT-US-982-5968.

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals with large B-cell lymphoma, including Diffuse large B-cell lymphoma (DLBCL) not otherwise specified, Primary mediastinal large B-cell lymphoma (PMBCL), High-grade B-cell lymphoma (HGBL), and DLBCL arising from Follicular lymphoma (FL)
* Individuals must have relapsed disease after 2 or more lines of systemic therapy, or chemorefractory disease defined as the following:

  * No response to first-line therapy, including the following:

    * Progressive disease (PD) as best response to first therapy
    * Stable disease (SD) as best response after ≥ 4 cycles of first-line therapy (eg, 4 cycles of rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone (R-CHOP)), with SD duration no longer than 6 months from the last dose of therapy
  * No response to ≥ 2 lines of therapy, including the following:

    * PD as best response to most recent therapy
    * SD as best response after ≥ 2 cycles of last line of therapy
* Individuals must have received adequate prior therapy including at a minimum:

  * Anti-CD20 monoclonal antibody unless investigator determines that tumor is CD20 negative, and
  * An anthracycline-containing chemotherapy regimen
* At least 1 measurable lesion according to the International Working Group Lugano Classification. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy.
* Magnetic resonance imaging of the brain showing no evidence of central nervous system (CNS) lymphoma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Individuals with a known medical history of tuberculosis or a risk for tuberculosis exposure require negative tuberculosis testing by either tuberculin skin test or interferon gamma release assay.
* Adequate bone marrow function as evidenced by:

  * Absolute neutrophil count ≥ 1000/μL
  * Platelets ≥ 75,000/μL
  * Absolute lymphocyte count ≥ 100/μL
* Adequate renal, hepatic, cardiac, and pulmonary function as evidenced by:

  * Creatinine clearance (Cockcroft-Gault) ≥ 60 mL/min
  * Serum alanine aminotransferase or aspartate aminotransferase ≤ 2.5 upper limit of normal
  * Total bilirubin ≤ 1.5 mg/dL, except in individuals with Gilbert's Syndrome
  * Cardiac ejection fraction ≥ 50% with no evidence of clinically significant pericardial effusion as determined by echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings
  * No clinically significant pleural effusion
  * Baseline oxygen saturation > 92% on room air

Key Exclusion Criteria:

* History of Richter's transformation of chronic lymphocytic leukemia
* Autologous stem cell transplant (SCT) within 6 weeks of planned axicabtagene ciloleucel infusion
* History of allogeneic stem cell transplantation
* Prior CD19 targeted therapy or prior CAR T cell therapy
* History of pulmonary alveolar proteinosis (PAP)
* History of severe, immediate hypersensitivity reaction attributed to aminoglycosides
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B (HBsAg positive) or hepatitis C (HCV) (anti-HCV positive) infection. A history of hepatitis B or hepatitis C infection is permitted if the viral load is undetectable per quantitative polymerase chain reaction (PCR) and/or nucleic acid testing.
* Individuals with detectable Cerebrospinal fluid (CSF) malignant cells, or brain metastases, or with a history of CNS lymphoma, CSF malignant cells or brain metastases
* History or presence of CNS disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2022-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (10):
- United States (10):
  - Stanford University, Palo Alto, California
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Evanston, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, New York-Presbyterian Hospital, New York, New York
  - Levine Cancer Center, Charlotte, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy/
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy/

REFERENCES:
- [Background] Kenderian, S. S., Oluwole, O. O., Mccarthy, P. L., Reshef, R., Shiraz, P., Ahmed, O., Le Gall, J., Nahas, M., Tang, L. And Neelapu, S. S. Zuma-19: A Phase 1/2 Multicenter Study of Lenzilumab Use With Axicabtagene Ciloleucel (Axi-Cel) In Patients (Pts) With Relapsed Or Refractory Large B Cell Lymphoma (R/R Lbcl). Blood 136(Supplement 1): 6-7, (2020). Conference Proceedings.
- [Background] Olalekan O. Oluwole, MBBS, Saad S. Kenderian, MD, Parveen Shiraz, MD, Reem Karmali, MD, MSc, Ran Reshef, MD, MSc, Philip L. McCarthy, MD, Nilanjan Ghosh, MD, PhD, Aleksandr Lazaryan, MD, PhD, MPH, Simone Filosto, PhD, Soumya Poddar, PhD, Daqin Mao, PhD, Andrew Peng, MS, Adrian Kilcoyne, MD, MPH, Myrna Nahas, MD, Sattva S. Neelapu, MD. A Phase 1/2 Study of Axicabtagene Ciloleucel Plus Lenzilumab in Patients With Relapsed or Refractory Large B-Cell Lymphoma. American Society of Hemotology; Dec 10-13, 2022; New Orleans, LA. Abstract 4635
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KT-US-471-0119

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States.
Pre-assignment Details: 9 participants were screened. The study was terminated earlier than planned, and thus the study did not proceed to Phase 2.
Groups:
- Phase 1/Cohort 1: Participants received 500 mg/m^2 cyclophosphamide intravenously (IV) and 30 mg/m^2/day fludarabine IV lymphodepleting chemotherapy followed by sequenced therapy of 600 mg lenzilumab IV and axicabtagene ciloleucel IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg on Day 0 to determine a recommended Phase 2 dose (RP2D) of lenzilumab. For participants weighing greater than 100 kg, a maximum flat dose of 2 x 10^8 anti-CD19 CAR T cells was administered.
- Phase 1/Cohort 2: Participants received 500 mg/m^2 cyclophosphamide IV and 30 mg/m^2/day fludarabine IV lymphodepleting chemotherapy followed by sequenced therapy of 1800 mg lenzilumab IV and axicabtagene ciloleucel IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg on Day 0 to determine RP2D of lenzilumab. For participants weighing greater than 100 kg, a maximum flat dose of 2 x 10^8 anti-CD19 CAR T cells was administered.
Period: Overall Study
Arm/Group | Phase 1/Cohort 1 | Phase 1/Cohort 2
Started | 3 | 3
Completed | 0 | 0
Not Completed | 3 | 3
Not completed — Death | 2 | 2
Not completed — Rolled over to long-term follow-up study after study terminated | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants treated with any dose of axicabtagene ciloleucel and/or any dose of lenzilumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1/Cohort 1 | Phase 1/Cohort 2 | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (15.7) | 65 (10.2) | 64 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Percentage of Participants Experiencing Adverse Events (AEs) Defined as Dose Limiting Toxicities (DLTs) Related to Sequenced Therapy With Lenzilumab and Axicabtagene
Description: A DLT was defined as the following sequenced therapy-related events with onset within the first 28 days following lenzilumab and axicabtagene ciloleucel infusions:
  * Grade 4 neutropenia lasting longer than 21 days from the day of cell transfer
  * Grade 4 thrombocytopenia lasting longer than 28 days from the day of cell transfer
  * Any sequenced therapy-related AE requiring intubation, including Grade 4 encephalopathy requiring intubation for airway protection
  * Any sequenced therapy-related Grade 5 event
Time Frame: First infusion of lenzilumab and axicabtagene ciloleucel up to 28 days.
Population: DLT evaluable set included all participants treated in the Phase 1 dosing cohort who received the target dose of lenzilumab and axicabtagene ciloleucel and were followed for at least 28 days after the anti-CD19 CAR T cell infusion or who received a dose of lenzilumab lower than target dose for that cohort and experienced a DLT during the 28-day after the anti-CD19 CAR T cell infusion.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1/Cohort 1 | Phase 1/Cohort 2
Number analyzed (Participants) | 3 | 3
percentage of participants | 0 | 0

2. Primary Outcome: Phase 2: Percentage of Participants Experiencing Grade 2 or Higher Neurologic Events Within 28 Days of Axicabtagene Ciloleucel Administration
Time Frame: Up to 28 days
Population: Due to early termination of study, Phase 2 of the study was not conducted.
Groups:
- Phase 2: Participants were to received 500 mg/m^2 cyclophosphamide IV and 30 mg/m^2/day fludarabine IV lymphodepleting chemotherapy followed by sequenced therapy of lenzilumab IV (at RP2D, dose selected based on Phase 1) and axicabtagene ciloleucel IV at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg but the study was terminated before proceeding to Phase 2.
Arm/Group | Phase 2
Number analyzed (Participants) | 0

3. Secondary Outcome: Phase 1 and Phase 2: Percentage of Participants Experiencing Adverse Events
Time Frame: Enrollment through 3 months after lenzilumab and axicabtagene ciloleucel infusion.
Population: For Phase 1, participants in the Safety Analysis Set were analyzed. Due to early termination of study, Phase 2 of the study was not conducted.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1/Cohort 1 | Phase 1/Cohort 2
Number analyzed (Participants) | 3 | 3
percentage of participants | 100 | 100

4. Secondary Outcome: Phase 1 and Phase 2: Percentage of Participants Experiencing Serious Adverse Events
Time Frame: Enrollment through 3 months after lenzilumab and axicabtagene ciloleucel infusion.
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1/Cohort 1 | Phase 1/Cohort 2
Number analyzed (Participants) | 3 | 3
percentage of participants | 67 | 100

5. Secondary Outcome: Phase 1 and Phase 2: Percentage of Participants Experiencing Cytokine Release Syndrome
Time Frame: Enrollment through 12 months after lenzilumab and axicabtagene ciloleucel infusion or until disease progression, whichever occurred first.
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1/Cohort 1 | Phase 1/Cohort 2
Number analyzed (Participants) | 3 | 3
percentage of participants | 67 | 67

6. Secondary Outcome: Phase 1 and Phase 2: Percentage of Participants Experiencing Neurologic Events
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1/Cohort 1 | Phase 1/Cohort 2
Number analyzed (Participants) | 3 | 3
percentage of participants | 100 | 67

7. Secondary Outcome: Phase 1 and Phase 2: Complete Response (CR) Rate Per Internal Working Group (IWG) Lugano Classification as Determined by the Study Investigators
Description: CR rate: percentage of participants with CR (CMR;CRR). CMR: positron emission tomography(PET)5-point scale(5PS) scores of 1(no uptake above background), 2(uptake ≤ mediastinum), 3(uptake > mediastinum but ≤ liver) with/without a residual mass); no new sites; and no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow. CRR: target nodes/nodal masses regressed to ≤ 1.5 cm in longest transverse diameter (LDi) of a lesion; no extra lymphatic sites; absent non-measured lesion;organ enlargement regress to normal; no new sites; and bone marrow normal by morphology.
Time Frame: First infusion date axicabtagene ciloleucel to data cut off date of 09 May 2022 (maximum duration: 22.3 months).
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1/Cohort 1 | Phase 1/Cohort 2
Number analyzed (Participants) | 3 | 3
percentage of participants | 67 [9 to 99] | 67 [9 to 99]

8. Secondary Outcome: Phase 1 and Phase 2: Objective Response Rate (ORR) Per IWG Lugano Classification as Determined by Study Investigators
Description: ORR: Percentage of participants with CR(CMR;CRR) or PR(partial metabolic response(PMR);partial radiologic response (PRR)).CMR:PET 5PS scores of 1,2,3 with/without a residual mass;no new sites;no evidence of FDG-avid disease in bone marrow.CRR:target nodes/nodal masses regressed to ≤ 1.5 cm in LDi of a lesion;no extra lymphatic sites;absent non-measured lesion;organ enlargement regress to normal;no new sites;bone marrow normal by morphology.PMR:5PS scores of 4(uptake moderately higher than liver),or 5(uptake markedly higher than liver and/or new lesions),with reduced uptake compared to baseline and residual masses of any size;no new sites;residual update > update in normal bone marrow but reduced compared with baseline.PRR:≥ 50% decrease in sum of the product of perpendicular diameters of up to 6 target measurable nodes and extranodal sites;absent/normal, regressed, but no increase of nonmeasured lesions;spleen regressed by > 50% in length beyond normal;no new sites.
Time Frame: First infusion date axicabtagene ciloleucel to data cut off date of 09 May 2022 (maximum duration: 22.3 months).
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1/Cohort 1 | Phase 1/Cohort 2
Number analyzed (Participants) | 3 | 3
percentage of participants | 67 [9 to 99] | 100 [29 to 100]

9. Secondary Outcome: Phase 1 and Phase 2: Duration of Response (DOR) in Participants Who Experience an Objective Response Per IWG Lugano Classification as Determined by Study Investigators
Description: DOR is defined only for participants who experience an objective response after axicabtagene ciloleucel infusion and is the time from the first objective response to disease progression or death from any cause. Objective response is defined in outcome measure (OM) 7.
Time Frame: First infusion date axicabtagene ciloleucel to data cut off date of 09 May 2022 (maximum duration: 22.3 months).
Population: For Phase 1, participants in the Safety Analysis Set with available data were analyzed. Due to early termination of study, Phase 2 of the study was not conducted.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1/Cohort 1 | Phase 1/Cohort 2
Number analyzed (Participants) | 2 | 3
Months | 9.9 [NA to NA] — The lower and upper limit of Confidence Interval (CI) was not estimable due to insufficient number of participants with an event. | 12.1 [2.7 to NA] — The upper limit of CI was not estimable due to insufficient number of participants with an event.

10. Secondary Outcome: Phase 1 and Phase 2: Progression-Free Survival (PFS) Per IWG Lugano Classification as Determined by Study Investigators
Description: PFS is defined as the time from the axicabtagene ciloleucel infusion date to the date of disease progression per Lugano classification or death from any cause.
Time Frame: First infusion date axicabtagene ciloleucel to data cut off date of 09 May 2022 (maximum duration: 22.3 months).
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1/Cohort 1 | Phase 1/Cohort 2
Number analyzed (Participants) | 3 | 3
Months | 10.8 [0.9 to NA] — The upper limit of Confidence Interval (CI) was not estimable due to insufficient number of participants with an event. | 13.0 [3.6 to NA] — The upper limit of CI was not estimable due to insufficient number of participants with an event.

11. Secondary Outcome: Phase 1 and Phase 2: Overall Survival (OS)
Description: OS is defined as the time from axicabtagene ciloleucel infusion to the date of death.
Time Frame: First infusion date axicabtagene ciloleucel to data cut off date of 09 May 2022 (maximum duration: 22.3 months).
Population: Phase 1, participants in the Safety Analysis Set were analyzed. Due to early termination of study, Phase 2 of the study was not conducted.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1/Cohort 1 | Phase 1/Cohort 2
Number analyzed (Participants) | 3 | 3
Months | 10.8 [4.6 to NA] — The upper limit of Confidence Interval (CI) was not estimable due to insufficient number of participants with an event. | 13.0 [3.6 to NA] — The upper limit of CI was not estimable due to insufficient number of participants with an event.

12. Secondary Outcome: Phase 1 and Phase 2: Pharmacodynamics: Peak Serum Level of CXCL10, Granzyme B, IFN-gamma, IL-1 RA, IL-2, IL-6, IL-8, TNF Alpha, GM-CSF, and MCP-1
Description: Peak is defined as the maximum post-baseline level of the analyte from baseline to Week 4.
Time Frame: Baseline up to Week 4
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Phase 1/Cohort 1 | Phase 1/Cohort 2
Number analyzed (Participants) | 3 | 3
pg/mL
  CXCL10 | 2000.00 [1474.50 to 2000.00] | 809.40 [448.60 to 1298.10]
  Granzyme B | 14.50 [9.20 to 44.20] | 11.80 [2.60 to 17.80]
  IFN-gamma | 1238.30 [90.60 to 1426.00] | 45.70 [7.50 to 151.50]
  IL-1 RA | 4984.00 [4038.00 to 6187.00] | 919.00 [701.00 to 1099.00]
  IL-2 | 11.80 [6.30 to 22.70] | 18.20 [2.50 to 21.10]
  IL-6 | 22.50 [8.00 to 976.00] | 13.10 [3.00 to 15.40]
  IL-8 | 56.70 [12.90 to 75.70] | 31.50 [15.40 to 39.90]
  TNF alpha | 5.50 [3.40 to 16.50] | 3.00 [1.70 to 3.30]
  GM-CSF | 1.90 [1.90 to 1.90] | 1.90 [1.90 to 1.90]
  MCP-1 | 1178.10 [1007.00 to 1300.00] | 866.80 [589.90 to 968.90]

13. Secondary Outcome: Phase 1 and Phase 2: Axicabtagene Ciloleucel Pharmacokinetics: Peak Level of Anti-CD19 CAR T Cells in Blood
Description: Peak is defined as the maximum number of CAR T cells in blood measured after the axicabtagene ciloleucel infusion.
Time Frame: Baseline up to Month 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Phase 1/Cohort 1 | Phase 1/Cohort 2
Number analyzed (Participants) | 3 | 3
cells/μL | 74.28 (97.60) | 20.35 (15.12)

ADVERSE EVENTS:
Time Frame: Adverse Events: Enrollment through 3 months after lenzilumab and axicabtagene ciloleucel infusion. All-Cause Mortality: Enrollment up to 22.5 months
Description: Adverse Events and All-Cause Mortality: The Safety Analysis Set included all participants treated with any dose of axicabtagene ciloleucel and/or any dose of lenzilumab.
Arm/Group | Phase 1/Cohort 1 | Phase 1/Cohort 2
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1/Cohort 1 (N=3) | Phase 1/Cohort 2 (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Covid-19 (Infections and infestations) | 0 | 1
Covid-19 pneumonia (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 2
Agitation (Psychiatric disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1/Cohort 1 (N=3) | Phase 1/Cohort 2 (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 2
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 2 | 1
Malaise (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 2
Tenderness (General disorders) | 0 | 1
Candida infection (Infections and infestations) | 1 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Diffuse large B-cell lymphoma refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Dysgraphia (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 2
Seizure (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 2
Confusional state (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT04314843/Prot_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT04314843/SAP_001.pdf
  • Statistical Analysis Plan: Translational Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT04314843/SAP_002.pdf